CLINICAL TRIAL: NCT07246655
Title: Effects of High-Intensity Inspiratory Muscle Training on Respiratory Muscle Strength, Balance, and Core Endurance in American Football Players
Brief Title: Inspiratory Muscle Training in American Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Namik Kemal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YeditepeU 312
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Inspiratory Muscle Training
Keywords: inspiratory muscle training; tackle football; core endurance; balance; performance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Inspiratory Muscle Training Group (Experimental): Inspiratory muscle training Team strength and conditioning training
  Interventions: Behavioral: High-Intensity Inspiratory Muscle Training
- Control Group (Active Comparator): Team strength and conditioning training
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: High-Intensity Inspiratory Muscle Training — Participants in the IMT Group will perform an 8-week high-intensity inspiratory muscle training protocol in addition to their routine team-based strength and conditioning program. Training loads will be individualized based on each athlete's maximal inspiratory pressure (MIP) and set at approximately 80% of MIP. Loads will be reassessed every two weeks, and the resistance will be adjusted to maintain the prescribed intensity.
  Arms: High-Intensity Inspiratory Muscle Training Group
Behavioral: Control Group — Participants in the Control Group will continue their standard team-based strength, conditioning, and field training sessions throughout the 8-week study period. They will not receive inspiratory muscle training or any additional respiratory intervention.
  Arms: Control Group

SUMMARY:
The aim of the randomized controlled study is to investigate the effects of high-intensity inspiratory muscle training on respiratory strength, balance, and core endurance in American Football (Tackle Football) athletes.

DETAILED DESCRIPTION:
After completing baseline assessments, participants will be randomly assigned to either the High-Intensity Inspiratory Muscle Training group (IMT Group) or the Control Group (CG) using simple randomization procedures.

All athletes in both groups will continue their regular team-based strength and conditioning routines throughout the 8-week study period. Participants in the IMT Group will additionally perform a high-intensity inspiratory muscle training protocol three times per week, with training loads set at approximately 80% of each athlete's measured maximal inspiratory pressure (MIP). Training intensity will be reassessed bi-weekly and adjusted according to updated MIP values to ensure that the prescribed load is maintained throughout the intervention. The Control Group will not receive inspiratory muscle training and will perform only their routine training program.

All athletes will be evaluated at baseline and at the end of the 8-week intervention. Outcome measures will include respiratory muscle strength (MIP/MEP), dynamic and static balance performance, core muscle endurance (McGill core endurance tests), and sport-specific performance parameters relevant to American football. Assessments will be carried out by the same researcher to minimize inter-rater variability, and all training sessions will be supervised to ensure protocol adherence.

Data will be collected and recorded systematically at both time points, and all procedures will follow established ATS/ERS guidelines for respiratory muscle testing and standard sports science assessment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified male American football athletes
* Ages 18 to 35 years
* Actively participating in team-based training at the time of study enrollment
* Minimum 1 year of organized American football training experience
* Able to perform high-intensity inspiratory muscle training (IMT)
* No history of acute respiratory infection in the past 4 weeks
* Voluntary agreement to participate and ability to provide informed consent

Exclusion Criteria:

* Acute or chronic respiratory disease (e.g., uncontrolled asthma, COPD)
* History of major cardiovascular, neurological, or musculoskeletal disorders affecting performance
* Current rib, spine, abdominal, or core muscle injury
* Diagnosed pulmonary hypertension or unstable cardiac conditions
* Recent surgery (within the past 3 months)
* Inability to correctly perform inspiratory muscle training (IMT) device technique
* Participation in another interventional study within the last 30 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be self-identified male American football athletes actively participating in team training.
Enrollment: 24 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure test | Baseline and after 8 weeks of training
  Maximal inspiratory pressure (MIP) will be measured at the mouth using a handheld pressure manometer in accordance with ATS/ERS recommendations. Participants will perform at least three maximal inspiratory efforts from residual volume, and the highest reproducible value will be recorded in cmH₂O.
Maximal Expiratory Pressure (MEP) | Baseline and after 8 weeks of training
  Maximal expiratory pressure (MEP) will be assessed with a handheld pressure manometer according to ATS/ERS standards. Participants will perform at least three maximal expiratory efforts from total lung capacity, and the highest reproducible value will be recorded in cmH₂O.

SECONDARY OUTCOMES:
Core muscle endurance | Baseline and after 8 weeks of training
  Core muscle endurance will be evaluated using the McGill core endurance tests (trunk flexor endurance, trunk extensor endurance, and right/left lateral plank endurance). During each test, participants will maintain the required test position as long as possible, and endurance time will be recorded in seconds.
Balance Performance (Static and Dynamic) | Baseline and after 8 weeks
  Balance performance will be evaluated using a computerized balance analysis system. Standardized static and dynamic balance tasks will be performed, and stability indices/output parameters provided by the system will be recorded.
Vertical Jump Height | Baseline and after 8 weeks
  Vertical jump performance will be assessed using a validated force platform or jump measurement device. Participants will perform three maximal countermovement jumps with hands on hips, and the highest reproducible jump height will be recorded in centimeters.
Isometric Leg Strength | Baseline and after 8 weeks
  Isometric leg strength will be measured using an isometric dynamometer (e.g., Takei Back and Leg Dynamometer). Participants will perform three maximal isometric leg extension or leg-back pulling efforts following standardized testing instructions. The highest reproducible value (kg or Newtons) will be recorded.
Yo-Yo Intermittent Recovery Test Level 1 Performance (Yo-Yo IR1) | Baseline and after 8 weeks
  The Yo-Yo Intermittent Recovery Test Level 1 will be administered following the standard protocol. Total distance completed (meters) before volitional exhaustion or failure to meet audio cues will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Develi, PhD., Principal Investigator — Yeditepe University
Locations (1):
- Tekirdağ Namık Kemal Univercity, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is a graduate thesis project involving a limited sample of athletes, and data cannot be publicly released to protect participant privacy.